CLINICAL TRIAL: NCT05369429
Title: My Wellbeing Guide, Technology Facilitated Behavioral Intervention for Depression Among Diverse Patients in Ambulatory Oncology
Brief Title: My Wellbeing Guide: a Novel Tool for Managing Stress and Improving Quality of Life
Acronym: R37
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Miami (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Betina Yanez, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00213537; 1R37CA255875-01 (NIH)
Record Dates: First submitted 2022-04-29; First posted 2022-05-11 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Anxiety; Depressive Symptoms
Keywords: eHealth; Wellbeing
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention includes cognitive behavioral therapy management strategies for health-related stress in the form of animated videos, interactive activities, and written content. The intervention will be delivered via an online application over an 7-week period. Intervention participants will also complete four assessments: baseline (at the beginning of the research study), post-intervention (7 weeks after baseline), a 6-month follow-up, and a 12-month follow up.
  Interventions: Behavioral: My Wellbeing Guide
- Control (No Intervention): The control application will provide links to helpful resources for patients with cancer, such as the contact information for cancer support services at Northwestern University and the University of Miami, and the link to the National Cancer Institute website, and the American Cancer Society website. Control participants will also complete four assessments: baseline (at the beginning of the research study), post-intervention (7 weeks after baseline), a 6-month follow-up, and a 12-month follow up.

INTERVENTIONS:
Behavioral: My Wellbeing Guide — The intervention includes cognitive behavioral therapy management strategies for health-related stress in the form of animated videos, interactive activities, and written content. The intervention will be delivered via an online application over an 7-week period. Intervention participants will also complete four assessments: baseline (at the beginning of the research study), post-intervention (7 weeks after baseline), a 6-month follow-up, and a 12-month follow up.
  Arms: Intervention

SUMMARY:
The purpose of this study is to examine the implementation and effectiveness of the psychosocial eHealth intervention, My Wellbeing Guide, on the proposed primary outcome, depressive symptoms, in patients diagnosed with cancer who receive care at Northwestern Medicine and the University of Miami Health System. Eligible patients will be directly contacted by the study team for recruitment.

The intervention includes cognitive behavioral therapy management strategies for health-related stress in the form of animated videos, interactive activities, and written content. The intervention will be delivered via an online application over an 7-week period. Intervention participants will also complete four assessments: baseline (at the beginning of the research study), post-intervention (7 weeks after baseline), a 6-month follow-up, and a 12-month follow up.

Participants are randomized into either an intervention application (described above) or a control application (which will provide links to helpful resources for patients with cancer, such as the contact information for cancer support services at Northwestern University and the University of Miami, and the link to the National Cancer Institute website, and the American Cancer Society website.) Control participants will also complete four assessments: baseline (at the beginning of the research study), post-intervention (7 weeks after baseline), a 6-month follow-up, and a 12-month follow up.

DETAILED DESCRIPTION:
Depression is one of the most common psychological comorbidities experienced throughout the cancer continuum. Elevated depressive symptoms in oncology patients is a major concern as unmanaged depressive symptoms in cancer patients is associated with poor health-related quality of life (HRQoL), poor adherence to cancer treatments, delayed return to work and baseline function, greater emergency department visits, and higher all-cause mortality. Behavioral interventions for the management of depression are efficacious, but scalability and implementation of these evidence-based interventions in oncology is limited. Health information technologies (HIT) provide an ideal opportunity to expedite the administration, scoring, and interpretation of depression screening with well-validated, brief and precise measurement tools that can capture actionable data to screen for depression, and deliver pragmatic and scalable evidence-based behavioral interventions that are proven to reduce depressive symptomatology across various other populations.

The study takes place across two distinct health systems in two major metropolitan areas-Chicago and Miami (Northwestern Medicine and University of Miami Health System). While across the two health systems (NM and UHealth), patients already receive EHR-delivered assessments that are linked to EPIC and real-time alerts sent to supportive oncology for patients with moderately to severely elevated symptoms, a lacking component is the integration of an evidence-based, HIT management program for elevated depressive symptoms.

The investigators will evaluate the effectiveness and the implementation of an evidence-based HIT behavioral treatment for cancer patients with elevated depressive symptoms. This HIT treatment combines systematic, electronic health record-integrated screening for depressive symptoms with an individually-tailored HIT interventions to address gaps in the treatment of depression among cancer patients. The investigators' specific aims are as follows:

Aim 1a. To further develop and refine My Wellbeing Guide, a web-based platform to optimize management of elevated depressive symptoms in ambulatory oncology in two large health systems.

Aim 1b. To establish the effectiveness of My Wellbeing Guide on depressive symptoms (i.e., primary outcome) and anxiety, HRQoL, and health services utilization (i.e. secondary outcomes), and putative mechanisms of action/mediators (e.g., self -efficacy) of My Wellbeing Guide on study outcomes compared to usual care.

Aim 1c. To evaluate the process of implementing My Wellbeing Guide and its impact on patient and system-level outcomes through electronic health record (EHR) extractions of Aim 1b patients, and through clinician, and hospital administrator interviews.

Aim 2. To identify facilitators and barriers to wide-scale implementation and expansion of My Wellbeing Guide through interviews and focus groups with stakeholders (clinicians, hospital administrators, and patients who participated in My Wellbeing Guide).

ELIGIBILITY:
Inclusion Criteria:

a) having been reached out to by the study team for recruitment; (b) planned treatment and follow-up within the NM or UHealth healthcare system; (c) ≥ 18 years of age; (d) medical chart confirmed diagnosis of a solid or hematological malignancy; (e) elevated depressive symptoms on the PROMIS CAT (score > or = 55) within the last 3 months; (f) access to the internet; (g) willingness to be randomized; (h) able to read English or Spanish; (i) patients must have signed informed consent prior to registration on study

Exclusion Criteria:

Note: The investigators will not include any vulnerable populations in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6516 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms will be evaluated with the Patient-Reported Outcomes Measurement Information System Depression | T1 (prior to starting intervention), T2 (7 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post-intervention)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression questionnaire is a previously validated patient-report measure of depressive symptoms in the last seven days. Scores generally range from 20 - 80, with higher scores indicating a patient is reporting more severe levels of depression.

SECONDARY OUTCOMES:
Change in anxiety will be evaluated with the Patient-Reported Outcomes Measurement Information System Anxiety | T1 (prior to starting intervention), T2 (7 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post-intervention)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety questionnaire is a previously validated patient-report measure of symptoms of anxiety in the last seven days. Scores generally range from 20 - 80, with higher scores indicating a patient is reporting more severe levels of anxiety.
Change in Health Related Quality of Life will be evaluated with The Functional Assessment of Cancer Therapy - General - 7 item version (FACT-G7) | T1 (prior to starting intervention), T2 (7 weeks post intervention), T3 (6 months post-intervention), T4 (12 months post-intervention)
  The Functional Assessment of Cancer Therapy - General - 7 item version (FACT-G7) has been used extensively to measure Health Related Quality of Life (HRQoL). The FACT-G7assesses participant's wellbeing in physical, emotional, social, and functional concerns in the last seven days using a five-point response scale. Scores range from 0-28, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Betina Yanez, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No